CLINICAL TRIAL: NCT02089516
Title: Activity Monitoring in Frail Elderly Patients. A Methods Comparison Study.
Brief Title: Activity Monitoring in Frail Elderly Patients
Status: Completed | Type: Observational
Sponsor: Medical Research Foundation, The Netherlands (Other)
Responsible Party: Principal Investigator, Henk Bilo, MD, MD PhD, Medical Research Foundation, The Netherlands
Other Study IDs: DynaPort I
Record Dates: First submitted 2014-03-14; First posted 2014-03-17 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Elderly
Keywords: Frailty; Accelerometry; Physical activity; validity
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Frail elderly: Measuring movement activity in frail elderly (GFI score ≥ 4) of 75 years and older using DynaPort.

SUMMARY:
The purpose of this stuydy is to assess the bias and repeatability of the DynaPort MicroMod in measuring movement / physical activity in frail elderly.

DETAILED DESCRIPTION:
Elderly subjects will be recruited from a residential-care complex in Zwolle, the Netherlands. All subjects will be asked to fill in the Groningen Frailty Index. We aim to select patients with varying GFI scores to ensure that we include patients with different degrees of frailty. The participating subjects will be asked to wear the DynaPort MicroMod during six hours. Two research employees will observe all activities of the participating subjects in their home environment. The participant will be instructed to act like it is a normal/usual day. Every 5 minutes the type of activity at that moment and movement intensity of the last 5 minutes (METs scale) is manually entered onto a case report form (CRF) by the two employees. The timing has to be exact in order to compare the data to the data of the DynaPort MicroMod. Type of activity is described as well as categorised into lying, sitting, standing or walking. Movement intensity is categorised according to a MET-value (Metabolic Equivalent of Task).

Sensitivity, specificity, and percentage of overall agreement will be calculated for each type of activity (standing, sitting, lying, walking) and for intensity. The primary analysis will be the comparison between walking and not walking (lying, sitting or standing). An overall agreement/sensitivity/specificity of 90% or higher is considered as sufficient agreement. The Bland and Altman method will also be used as multiple observations are recorded per patient, the limits of agreement will also be calculated with the Bland and Altman method for repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* Age: 75 years and older
* Frailty: GFI (Groningen Frailty Index) score ≥ 4

Exclusion Criteria:

* Living in a nursing-home

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Home-dwelling frail elderly (GFI score ≥ 4) of 75 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Type of movement: lying, sitting/standing or walking | up to six hours
  The participating subjects will be asked to wear the DynaPort MicroMod during six hours. Two research employees will observe all activities of the participating subjects in their home environment. Every 5 minutes the type of activity at that moment is manually entered onto a case report form (CRF) by the two research employees.

SECONDARY OUTCOMES:
Movement intensity (METs) | up to six hours
  The participating subjects will be asked to wear the DynaPort MicroMod during six hours. Two research employees will observe all activities of the participating subjects in their home environment. Every 5 minutes the movement intensity of the last 5 minutes (METs scale) is manually entered onto a case report form (CRF) by the two employees.

CONTACTS AND LOCATIONS:
Overall Officials: Kornelis van Hateren, MD PhD, Principal Investigator — Isala, diabetes centre
Locations (2):
- Netherlands (2):
  - Woonzorgcentrum De Wissel, Zwolle, Overijssel
  - Woonzorgcentrum Westenhage, Zwolle, Overijssel

REFERENCES:
- See also: Description of the DynaPort MicroMod used in this study — http://www.mcroberts.nl/